CLINICAL TRIAL: NCT07285031
Title: The Role of Histamines on Central Hemodynamics
Brief Title: Histamines and Central Hemodynamics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Neil Eves, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H25-01909
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Histamine; Exercise
Keywords: histamine; exercise; pulmonary blood flow; pulmonary function; femoral blood flow
MeSH Terms: conditions — Motor Activity | interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blockade + Exercise Bout (Experimental): Participants will ingest histamine H1 receptor blockade before performing an exercise bout.
  Interventions: Drug: Diphenhydramine hydrochloride; Other: Exercise Bout
- Placebo + Exercise Bout (Placebo Comparator): Participants will ingest a placebo before an exercise bout.
  Interventions: Other: Placebo; Other: Exercise Bout

INTERVENTIONS:
Drug: Diphenhydramine hydrochloride — H1 receptor antagonist: 50mg Diphenhydramine Hydrochloride
  Arms: Blockade + Exercise Bout
Other: Placebo — Placebo
  Arms: Placebo + Exercise Bout
Other: Exercise Bout — Participants will complete a total of three 5-minute high intensity exercise intervals, interspersed with 5-minute lower intensity exercise bouts (4 total), for a total of 35 minutes.

SUMMARY:
When we exercise, more blood flow goes to our muscles, challenging our blood vessels. Following exercise, blood flow remains elevated and seems to be the reason for many of the positive cardiovascular benefits that occur with exercise. When the actions of histamine, a molecule primarily known for its role in allergies, are blocked, there is an attenuated blood flow response following exercise. However, this effect has never been studied in the blood vessels that supply our lungs. The purpose of this study is to examine the effects of histamines on pulmonary hemodynamics following exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 19 - 39.
2. Willing to visit the lab on 3 separate occasions.

Exclusion Criteria:

1. Previously diagnosed heart condition,
2. Previously diagnosed lung condition (including asthma),
3. Previously diagnosed metabolic condition,
4. Currently smokers (cigarettes, electronic cigarettes, cannabis) or who have smoked within the last 3 months,
5. Resting blood pressure >140/90 mmHg,
6. Unable to obtain appropriate quality ultrasound images of the heart.,
7. Individuals without tricuspid regurgitation at rest to allow assessment of the primary outcome,
8. Pregnant or trying to become pregnant,
9. Breastfeeding,
10. Chronically take antihistamines (i.e. daily),
11. History of adverse reactions to antihistamines,
12. Never taken antihistamines previously,
13. Currently taking any medications (including oral contraceptives).

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Systolic pulmonary artery pressure | Pre-exercise and 10, 20, and 30-minutes post-exercise.
  The difference in systolic pulmonary artery pressure (measured as tricuspid regurgitation velocity using echocardiography) between the H1 blockade condition and the placebo condition.

SECONDARY OUTCOMES:
Tricuspid annular plane systolic displacement | Pre-exercise and 0, 10, 20, 30, 45, and 60 minutes post-exercise.
  The difference in tricuspid annular plane systolic displacement between the H1 receptor blockade condition and the placebo condition.
Right ventricular stroke volume | Pre-exercise and 0, 10, 20, 30, 45, and 60-minutes post-exercise.
  The difference in right ventricular stroke volume (measured using pulsed wave velocity of the right ventricular outflow tract velocity time integral) between the H1 receptor blockade condition and the placebo condition.
Femoral artery blood flow | Pre-exercise and 0, 10, 20, 30, 45, and 60-minutes post-exercise.
  The difference in femoral artery blood flow between the H1 receptor blockade condition and the placebo condition.
Mean arterial systemic pressure | Pre-exercise and 0, 10, 20, 30, 45, and 60-minutes post-exercise.
  The difference in mean arterial systemic pressure between the H1 receptor blockade condition and the placebo condition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided